CLINICAL TRIAL: NCT05166954
Title: Effect of Bariatric Surgery on Cardiac Function in Patients With Hypertension
Status: Recruiting | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-P2-254-02
Record Dates: First submitted 2021-12-12; First posted 2021-12-22 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Bariatric Surgery; Hypertension
Keywords: Cardiac Function; Echocardiography
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- LSG group: Laparoscopic sleeve gastrectomy (LSG) performed as a treatment for obesity
  Interventions: Procedure: LSG
- RYGB group: Laparoscopic Roux-en-Y gastric bypass performed as a treatment for obesity
  Interventions: Procedure: RYGB

INTERVENTIONS:
Procedure: LSG — Laparoscopic sleeve gastrectomy (LSG) together with medical treatment aiming the control of cardiovascular risks including hypertension, diabetes mellitus or dyslipidemia.
  Groups: LSG group
Procedure: RYGB — Roux-en-Y gastric bypass (LRYGB) together with medical treatment aiming the control of cardiovascular risks including hypertension, diabetes mellitus or dyslipidemia.
  Groups: RYGB group

SUMMARY:
The purpose of this study is to investigate the effect of bariatric surgery on cardiac function assessed by echocardiography in patients with hypertension.

DETAILED DESCRIPTION:
Obesity is the most common chronic metabolic disease worldwide, causing the increasing burden of cardiovascular risk factors such as hypertension, and affecting cardiac structure and function in the long term. Nowadays, bariatric surgery is regarded as the most effective approach for weight loss, and the only approach for reducing obesity-related cardiovascular events. However, the effect of different bariatric surgeries such as laparoscopic sleeve gastrectomy (LSG) or Roux-en-Y gastric bypass (RYGB) on cardiac function in patients with hypertension is still unclear. Therefore, the aim of this study was to evaluate the benefit of different bariatric surgeries on cardiac structure and function echocardiography in patients with hypertension.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old
* BMI>24kg/m2
* Bariatric surgery patients of Beijing Friendship Hospital
* History of hypertension and treated with ≥2 antihypertensive drugs for more than 4 weeks
* No major barriers to provide written consent

Exclusion Criteria:

* Secondary hypertension, except because of sleep apnea
* cardiovascular disease (myocardial infarction, heart failure, stroke or coronary revascularization) within 6 months
* Severe concomitant diseases (autoimmune disease, malignancy, late stage of liver diseases, respiratory diseases and digestive diseases)
* Unable to understand or comply with the study procedures

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Obese patients with hypertension
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes on left ventricular ejection fraction (LVEF) | 12 months
  Changes on LVEF in % assessed with the use of transthoracic echocardiography (TTE).

SECONDARY OUTCOMES:
Changes on left ventricular ejection fraction (LVEF) | 24 months
  Changes on LVEF in % assessed with the use of TTE.
Changes on left ventricular end-diastolic diameter (LVEDD) | 12 months
  Changes on LVEDD in mm assessed with the use of TTE.
Changes on left ventricular end-diastolic diameter (LVEDD) | 24 months
  Changes on LVEDD in mm assessed with the use of TTE.
Major adverse cardiac events | 12 months
  including all-cause mortality, cardiac death, acute myocardial infarction, stroke, heart failure, ventricular tachycardia or ventricular fibrillation requiring shock delivery.
Major adverse cardiac events | 24 months
  including all-cause mortality, cardiac death, acute myocardial infarction, stroke, heart failure, ventricular tachycardia or ventricular fibrillation requiring shock delivery.
Changes on number of antihypertensive drugs | 12 months
  Changes on of the total number of antihypertensive medications while maintaining office systolic and diastolic blood pressure <140 mm Hg and 90 mm Hg, respectively.
Changes on number of antihypertensive drugs | 24 months
  Changes on of the total number of antihypertensive medications while maintaining office systolic and diastolic blood pressure <140 mm Hg and 90 mm Hg, respectively.
Changes on blood pressure | 12 months
  Changes on systolic and blood pressure assessed with the use of 24-hour ABPM.
Changes on blood pressure | 24 months
  Changes on systolic and blood pressure assessed with the use of 24-hour ABPM.

CONTACTS AND LOCATIONS:
Overall Officials: Rongchong Huang, M.D., Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No